CLINICAL TRIAL: NCT00510887
Title: A Phase II Study of Bortezomib in Combination With Rituximab, Fludarabine, Mitoxantrone, and Dexamethasone (VR-FND) for Relapsed or Refractory Follicular Lymphoma
Brief Title: Bortezomib (Velcade) With Standard Chemotherapy for Relapsed or Refractory Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: Duke University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008487; 8785 (Other: DUMC old IRB number)
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: Lymphoma, Follicular
Keywords: follicular lymphoma; Velcade; VR-FND
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bortezomib; Rituximab; fludarabine; Mitoxantrone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VR-FND (Experimental): Bortezomib (VELCADER) 1.6 mg/m2 IV days 1 and 8 Rituximab 375 mg/m2 IV on day 1 Fludarabine 25 mg/m2 IV on days 1,2,3 Mitoxantrone 10 mg/m2 IV on day 2 Dexamethasone 20 mg orally on days 1,2,3,4,5 On day 1 the sequence of drug administration will be Bortezomib followed by Fludarabine followed by Rituximab.
  Each cycle will be repeated every 28 days for 8 cycles maximum.
  Interventions: Drug: Bortezomib; Drug: Rituximab; Drug: Fludarabine; Drug: Mitoxantrone; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.6 mg/m2 on days 1 and 8 of each 28-day cycle
  Other Names: Velcade
Drug: Rituximab — Rituximab 375 mg/m2 IV on day 1
Drug: Fludarabine — Fludarabine 25 mg/m2 IV on days 1,2,3
Drug: Mitoxantrone — Mitoxantrone 10 mg/m2 IV on day 2
  Other Names: Novantrone
Drug: Dexamethasone — Dexamethasone 20 mg orally on days 1,2,3,4,5

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of combining bortezomib (Velcade) with rituximab, fludarabine, mitoxantrone, and dexamethasone in treating patients with follicular cell lymphoma.

DETAILED DESCRIPTION:
This is a phase II study using the combination of bortezomib, rituximab, fludarabine, mitoxantrone and dexamethasone. The combination will given over a 28 day cycle. In addition each patient will receive Pneumocystis carinii Pneumonia (PCP) prophylaxis with Trimethoprim/sulfamethoxazole (TMP/Sulfa) or equivalent agent. On day 4 the physician has the option of starting granulocyte colony-stimulating factor (GCSF), granulocyte macrophage colony-stimulating factor (GMCSF), or pegylated GCSF.

All patients who receive at least one dose of the drug will be evaluated for toxicity. Patients will be treated with the agent for at least 2 cycles to be considered eligible for evaluation of response. The chemotherapy dosing will continue until there is evidence of disease progression, a second recurrence of unacceptable toxicity, or a maximum of 8 courses of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade 1-3 follicular lymphoma with persistent, relapsed, or refractory disease to at least one prior regimen.
* No prior bortezomib therapy.
* Voluntary written informed consent.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control.
* Male subject agrees to use an acceptable method for contraception for the duration of the study therapy.
* 18 years of age or older.
* aspartate aminotransferase (AST),alanine aminotransferase (ALT), total bilirubin < 3 times the upper limit of normal unless documented by the treating physician to be secondary to underlying lymphoma.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

* Platelet count of < 50,000 within 14 days before enrollment unless documented by the treating physician to be due to the disease.
* Absolute neutrophil count of < 1000 within 14 days before enrollment unless documented by the treating physician to be due to disease.
* Estimated or measured creatinine clearance of less than 30 ml/min within 14 days before enrollment.
* ≥Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia.
* Patient has hypersensitivity to boron, mannitol or any drug included in the current protocol.
* Female subject is pregnant or lactating.
* Received other investigational drugs for this disease within 14 days of enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Known HIV+ status.
* Cardiac ejection fraction less than 35% at study entry measured by echocardiogram, Multigated Acquisition (MUGA) or cardiac MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-01; Primary Completion 2012-11 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Rizzieri, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 14 subjects consented, 2 were screen failures so only 12 subjects received the study drug.
Groups:
- VR-FND: Bortezomib (VELCADE) 1.6 mg/m2 IV days 1 and 8 Rituximab 375 mg/m2 IV on day 1 Fludarabine 25 mg/m2 IV on days 1,2,3 Mitoxantrone 10 mg/m2 IV on day 2 Dexamethasone 20 mg orally on days 1,2,3,4,5 On day 1 the sequence of drug administration will be Bortezomib followed by Fludarabine followed by Rituximab.
  Each cycle will be repeated every 28 days for 8 cycles maximum.
  Bortezomib: Bortezomib 1.6 mg/m2 on days 1 and 8 of each 28-day cycle
  Rituximab: Rituximab 375 mg/m2 IV on day 1
  Fludarabine: Fludarabine 25 mg/m2 IV on days 1,2,3
  Mitoxantrone: Mitoxantrone 10 mg/m2 IV on day 2
  Dexamethasone: Dexamethasone 20 mg orally on days 1,2,3,4,5
Period: Overall Study
Arm/Group | VR-FND
Started | 12
Completed | 11
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All patients who were consented are included in the baseline analysis population.
Groups:
- VR-FND: Bortezomib (VELCADER) 1.6 mg/m2 IV days 1 and 8 Rituximab 375 mg/m2 IV on day 1 Fludarabine 25 mg/m2 IV on days 1,2,3 Mitoxantrone 10 mg/m2 IV on day 2 Dexamethasone 20 mg orally on days 1,2,3,4,5 On day 1 the sequence of drug administration will be Bortezomib followed by Fludarabine followed by Rituximab.
  Each cycle will be repeated every 28 days for 8 cycles maximum.
  Bortezomib: Bortezomib 1.6 mg/m2 on days 1 and 8 of each 28-day cycle
  Rituximab: Rituximab 375 mg/m2 IV on day 1
  Fludarabine: Fludarabine 25 mg/m2 IV on days 1,2,3
  Mitoxantrone: Mitoxantrone 10 mg/m2 IV on day 2
  Dexamethasone: Dexamethasone 20 mg orally on days 1,2,3,4,5
Arm/Group | VR-FND
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 72]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Complete and Partial Response
Description: * Complete Response: Complete disappearance of all detectable clinical and radiographic evidence of disease, disappearance of all disease-related symptoms and normalization of biochemical abnormalities (eg. LDH) definitely assignable to follicular lymphoma.
  * Partial Response requires the following:
    * greater than or equal to 50% decrease in the SPD of the 6 largest dominant nodes of nodal masses.
    * No increase in size of other nodes, liver, or spleen.
    * Splenic and hepatic nodes must regress by at least 50% in sum of the products (SPD).
    * Bone marrow assessment in irrelevant for determination of Partial Response since it is not measurable disease; however, if positive the type of cell should be reported.
    * No new lesions.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | VR-FND
Number analyzed (Participants) | 11
percentage of participants | 64

2. Secondary Outcome: Duration of Response
Description: Duration of response is measured from time of treatment to time of disease progression
Time Frame: up to 4 years
Measure: Mean (Full Range); unit: months
Arm/Group | VR-FND
Number analyzed (Participants) | 7
months | 16.47143 [3.4 to 43]

3. Secondary Outcome: Percentage of Subjects Experiencing Progression Free Survival
Description: Progression free survival is measured from treatment to progression or death, whichever comes first. Progressive disease is measured as: 50% or greater increase from nadir in the sum of the products (SPD) of any previously identified abnormal node and the appearance of any new lesions during or at the end of treatment.
Time Frame: up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | VR-FND
Number analyzed (Participants) | 11
percentage of participants | 17

4. Secondary Outcome: Percentage of Subjects Experiencing Overall Survival
Description: Overall survival is from the day of enrollment to date of death from any cause.
Time Frame: up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | VR-FND
Number analyzed (Participants) | 11
percentage of participants | 27

5. Secondary Outcome: Number of Participants With a Grade 3-4 Hematologic Toxicity.
Description: Before each drug dose, the patient will be evaluated for possible toxicities that may have occurred after the previous dose(s). Toxicities are to be assessed according to the NCI Common Toxicity Criteria (CTC).
Time Frame: up to 1 year
Measure: Number; unit: participants
Arm/Group | VR-FND
Number analyzed (Participants) | 11
participants | 7

6. Secondary Outcome: Number of Participants With Neuropathy, Any Grade
Description: as for outcome 5
Time Frame: up to 1 year
Measure: Number; unit: participants
Arm/Group | VR-FND
Number analyzed (Participants) | 11
participants | 6

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last dose of study drug
Description: All adverse events are reported whether or not they are considered attributable to the study treatment.
Arm/Group | VR-FND
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VR-FND (N=12)
Blood / Bone Marrow - Other (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (fever of unknown origin without documented infection) (Blood and lymphatic system disorders) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 8 (9)
Auditory / Ear (Ear and labyrinth disorders) | 1 (1)
Vision - blurred vision (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry mouth / salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Heartburn / dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis / Stomatitis (clinical exam) (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 8 (10)
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 (3)
Pain - Anus (Gastrointestinal disorders) | 1 (1)
Pain - Dental / teeth / peridontal (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (9)
Constitutional Symptoms - Other (General disorders) | 2 (2)
Edema: head and neck (General disorders) | 1 (1)
Edema: limb (General disorders) | 5 (5)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 10 (17)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2)
Pain - Chest / thorax NOS (General disorders) | 2 (2)
Rigors / chills (General disorders) | 3 (3)
Pain - Gallbladder (Hepatobiliary disorders) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
Infection with unknown ANC - Mucosa (Infections and infestations) | 1 (1)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
High Alkaline phosphatase (Investigations) | 4 (4)
High AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
High Creatinine (Investigations) | 3 (3)
Low Leukocytes (total WBC) (Investigations) | 10 (15)
Lymphopenia (Investigations) | 5 (5)
Metabolic / Laboratory - Other (Investigations) | 3 (4)
Low Neutrophils / granulocytes (ANC / AGC) (Investigations) | 7 (11)
Low Platelets (Investigations) | 9 (10)
Weight loss (Investigations) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 6 (10)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (9)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Uric Acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal - Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Back (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3 (4)
Dizziness (Nervous system disorders) | 3 (3)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 5 (5)
Pain - Head / headache (Nervous system disorders) | 3 (3)
Taste Alteration (dysgeusia) (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Mood Alteration - Agitation (Psychiatric disorders) | 1 (1)
Pain - Kidney (Renal and urinary disorders) | 1 (1)
Renal / Genitourinary - Other (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pain - Throat / pharynx / larynx (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Nail Changes (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae / purpura (hemorrhage / bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus / itching (Skin and subcutaneous tissue disorders) | 3 (3)
Rash / desquamation (Skin and subcutaneous tissue disorders) | 4 (6)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 5 (6)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes